CLINICAL TRIAL: NCT01286415
Title: Group Cognitive Processing Therapy for Combat-related PTSD
Brief Title: Group Cognitive Processing Therapy for Combat-related Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: STRONG STAR Multidisciplinary Research Consortium (Unknown); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Patricia Resick, Professor, Duke University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-08-2-0116
Record Dates: First submitted 2011-01-26; First posted 2011-01-31 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Cognitive Processing Therapy; combat; military; CPT; group therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Cognitive Processing Therapy-Cognitive Only (Experimental)
  Interventions: Behavioral: Group Cognitive Processing Therapy-Cognitive Only
- Group Present Centered Therapy (Active Comparator)
  Interventions: Behavioral: Group Present Centered Therapy

INTERVENTIONS:
Behavioral: Group Cognitive Processing Therapy-Cognitive Only — Cognitive Processing Therapy (CPT) is an evidence-based form of Cognitive Behavioral Therapy (CBT) used to treat PTSD. CPT is a 12-session manualized program that focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world. Sessions will be conducted twice weekly for six weeks; each session is 90 minutes.
  Arms: Group Cognitive Processing Therapy-Cognitive Only
Behavioral: Group Present Centered Therapy — Present Centered Therapy (PCT) is a supportive group intervention typically used within the Department of Veterans Affairs (VA) healthcare systems to address problems of veterans with PTSD (Rosen, et al., 2004). PCT focuses on problem-solving current difficulties that may be related to past traumatic events, but does not address specific memories or cognitions about the trauma. Sessions will be conducted twice weekly for 6 weeks; sessions are 90 minutes.
  Arms: Group Present Centered Therapy

SUMMARY:
The purpose of this study is to compare group-administered Cognitive Processing Therapy-Cognitive-only version (CPT-C), an evidence based treatment for posttraumatic stress disorder (PTSD), to Present Centered Therapy (PCT) in order to determine whether the results of CPT exceed those of receiving a therapy that focuses on current problems rather than past trauma in a group format.

DETAILED DESCRIPTION:
Estimates indicate that between 100,000 and 300,000 Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF) veterans are at significant risk for chronic post-traumatic stress disorder (PTSD), which can become a chronic disorder that impacts all areas of a person's life. PTSD treatment programs are being developed throughout the Department of Defense (DoD) and the Veterans Affairs (VA), but because of the large number of Service Members returning from deployment with PTSD, it is often necessary to provide psychotherapy in groups. Cognitive Processing Therapy (CPT), an evidence-based treatment for PTSD, was originally developed as a group-based intervention. However, group-based CPT treatment has never been systematically compared to other forms of group treatment. The public policy implications of the results of this trial are significant. If group treatment is found to be effective, then group treatment would be a more efficient and cost-effective therapy modality in most cases. The purpose of this study is to compare group-administered CPT-Cognitive-only version (CPT-C) to Present Centered Therapy (PCT) in order to determine whether the results of CPT exceed those of receiving a therapy that focuses on current problems rather than past trauma in a group format. One hundred (100) adult male and female active-duty OIF/OEF military personnel over 18 years of age will be enrolled into this study. Participants will be randomized to receive either group PCT or group CPT-C.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female active duty, activated Reservist, or activated National Guard OIF/OEF military personnel or OIF/OEF veterans seeking treatment for PTSD
* diagnosis of PTSD determined by a clinician-administered Posttraumatic Stress Scale (PSSI)
* person has experienced a Criterion A event that is a specific combat-related event or high magnitude operational experience that occurred during a military deployment in support of OIF/OEF. The diagnosis of PTSD may be indexed to that event or to another Criterion A event.
* be over the age of 18
* speak and read English
* be stable on any psychotropic medications they may be taking.

Exclusion Criteria:

* current suicide or homicide risk meriting crisis intervention
* active psychosis
* moderate to severe brain damage (as determined by the inability to comprehend the baseline screening questionnaires)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist-Stressor-specific Version (PCL-S) | Baseline, weekly during treatment, posttreatment, 6-month and 12-month follow-up
  PCL-S measures symptoms of posttraumatic stress disorder in response to a specific stressor.

SECONDARY OUTCOMES:
Beck Depression Inventory-II | Baseline, weekly during treatment, posttreatment, 6-month, and 12-month follow-up
  The BDI-II is one of the most widely used instruments for measuring the severity of depressive symptoms. It consists of 21 items that assess both affective and somatic symptoms related to depression and depressive disorders. Each item is composed of four statements that reflect symptom severity. The statements are scaled from 0 (no disturbance) to 3 (maximal disturbance). Scores on all items are summed to obtain a total severity score.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Resick, PhD, Principal Investigator — Duke University
Locations (1):
- Fort Hood Army Base, Fort Hood, Texas, United States

REFERENCES:
- [Background] Pruiksma KE, Taylor DJ, Wachen JS, Mintz J, Young-McCaughan S, Peterson AL, Yarvis JS, Borah EV, Dondanville KA, Litz BT, Hembree EA, Resick PA. Residual sleep disturbances following PTSD treatment in active duty military personnel. Psychol Trauma. 2016 Nov;8(6):697-701. doi: 10.1037/tra0000150. Epub 2016 May 30. PMID 27243567
- [Background] Dondanville KA, Blankenship AE, Molino A, Resick PA, Wachen JS, Mintz J, Yarvis JS, Litz BT, Borah EV, Roache JD, Young-McCaughan S, Hembree EA, Peterson AL; STRONG STAR Consortium. Qualitative examination of cognitive change during PTSD treatment for active duty service members. Behav Res Ther. 2016 Apr;79:1-6. doi: 10.1016/j.brat.2016.01.003. Epub 2016 Feb 4. PMID 26874683
- [Background] Bryan CJ, Clemans TA, Hernandez AM, Mintz J, Peterson AL, Yarvis JS, Resick PA; STRONG STAR Consortium. EVALUATING POTENTIAL IATROGENIC SUICIDE RISK IN TRAUMA-FOCUSED GROUP COGNITIVE BEHAVIORAL THERAPY FOR THE TREATMENT OF PTSD IN ACTIVE DUTY MILITARY PERSONNEL. Depress Anxiety. 2016 Jun;33(6):549-57. doi: 10.1002/da.22456. Epub 2015 Dec 4. PMID 26636426
- [Result] Resick PA, Wachen JS, Mintz J, Young-McCaughan S, Roache JD, Borah AM, Borah EV, Dondanville KA, Hembree EA, Litz BT, Peterson AL. A randomized clinical trial of group cognitive processing therapy compared with group present-centered therapy for PTSD among active duty military personnel. J Consult Clin Psychol. 2015 Dec;83(6):1058-1068. doi: 10.1037/ccp0000016. Epub 2015 May 4. PMID 25939018
- [Derived] Miles SR, Hale WJ, Mintz J, Wachen JS, Litz BT, Dondanville KA, Yarvis JS, Hembree EA, Young-McCaughan S, Peterson AL, Resick PA. Hyperarousal symptoms linger after successful PTSD treatment in active duty military. Psychol Trauma. 2023 Nov;15(8):1398-1405. doi: 10.1037/tra0001292. Epub 2022 Jul 28. PMID 35901423